CLINICAL TRIAL: NCT06188949
Title: A Randomized, Placebo-controlled, Feasibility Study to Evaluate Efficacy of Dietary Ingredient in Vitality & Metabolic Factors in Healthy Individuals
Brief Title: A Study to Evaluate Efficacy of Dietary Ingredient in Vitality and Metabolic Factors in Healthy Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vedic Lifesciences Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: EB/231101/DI/VMF
Record Dates: First submitted 2023-12-18; First posted 2024-01-03 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2024-04

CONDITIONS: Aging
MeSH Terms: interventions — Seeds

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled, double-blinded study
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dolichos biflorus (Horsegram) seed extract (Active Comparator): 1 capsule twice a day (Before breakfast & dinner)
  Interventions: Dietary Supplement: Dolichos biflorus (Horsegram) seed extract
- Carica papaya leaves extract (Active Comparator): 1 capsule twice a day (Before breakfast & dinner)
  Interventions: Dietary Supplement: Carica papaya leaves extract
- Placebo (MCC) (Placebo Comparator): 1 capsule twice a day (Before breakfast & dinner)
  Interventions: Dietary Supplement: Placebo (MCC)

INTERVENTIONS:
Dietary Supplement: Dolichos biflorus (Horsegram) seed extract — 1 capsule twice a day (Before breakfast & dinner)
  Arms: Dolichos biflorus (Horsegram) seed extract
Dietary Supplement: Carica papaya leaves extract — 1 capsule twice a day (Before breakfast & dinner)
  Arms: Carica papaya leaves extract
Dietary Supplement: Placebo (MCC) — 1 capsule twice a day (Before breakfast & dinner)
  Arms: Placebo (MCC)

SUMMARY:
The present study is a randomized, placebo-controlled, feasibility study to evaluate efficacy of dietary ingredients in vitality & metabolic factors in healthy individuals. Approximately 54 subjects aged between ≥ 40 and ≤ 60 years will be screened and 36 participants (12 in each arm) are to be randomized. Both the IP and placebo study arms will have 10 completed subjects in each arm after accounting for the screening failure and dropout/withdrawal rate of 30% and 17% respectively (Total 30 completers). The treatment duration for all the study subjects will be 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Physically active males and females aged ≥40 and ≤ 60 years
* Individuals with BMI ≥ 24.5 kg/m2 and ≤ 34.9 kg/m2
* Individuals with Fatigue Symptom Severity score ≥36 and ≤45
* Individuals with Perceived Stress score ≥20
* Having at least 2 of the following five metabolic risk factors:

  1. Waist circumference: Men: ≥ 102 cm (40.15 inches); Women ≥88 cm (34.65 inches)
  2. Triglycerides >150 mg/dL
  3. Systolic Blood pressure (SBP) ≥130 mm Hg and/or Diastolic Blood pressure (DBP) ≥85 mm Hg
  4. Fasting blood glucose ≥ 125 mg/ dl
  5. HDL level: Men: < 40 mg/dL; Women: < 50 mg/dL
* Individuals willing to provide signed Consent

Exclusion Criteria:

* Individuals on strict vegetarian diet.
* Individuals with fasting blood sugar ≥160 mg/dl
* Individuals currently hospitalized or planned for admission Individuals
* Individuals currently undergoing treatment with any other drugs such as insulin, corticoids, and non-steroidal anti-inflammatory drugs for more than 15 days.
* Individuals undergoing treatment of chemotherapy and/or suffering from AIDS, hepatitis, pregnancy are precluded from the study.
* Individuals undergoing chemotherapy
* Individuals suffering from AIDS, hepatitis.
* Individuals allergic to components of this nutraceutical formulations.
* Use of medications in the last 2 weeks prior to the pre-baseline period. This does not include birth control pills or standard multi-vitamin/mineral supplements.
* Daily use of NSAIDs in the last 3 months or incidental use in the last 2 weeks prior to screening.
* Abnormal Thyroid Stimulating Hormone (TSH) value which is < 0.40 or > 4.50 μIU/mL.
* Diagnosed cases of Type II Diabetes Mellitus with medication
* Hypertensive defined as SBP ≥ 160 mm Hg and/or DBP ≥ 100 mm Hg
* Individuals taking anti-hypertensive
* Individuals with dyslipidemia on medication
* Females in peri-menopausal state (Irregular menstrual period in last 6 months).
* Females on Hormone Replacement Therapy
* Individuals with a history of or complications from inflammatory conditions.
* Use of another investigational product within 3 months of the screening visit
* Individuals with a history of or complications from malignant tumors
* History of any significant neurological and psychiatric condition which may affect the participation and inference of the study's end points.
* Use of recreational drugs (such as cocaine, methamphetamine, marijuana, etc.)/Nicotine dependence.
* High-risk drinking as defined by consumption of 4 or more alcohol containing beverages on any day or 8 or more alcohol containing beverages per week for women and 5 or more alcohol containing beverages on any day or 15 or more alcohol containing beverages per week for men.
* Females who are pregnant/planning to be pregnant/lactating or taking any oral contraceptives.
* Any condition that could, in the opinion of the investigator, preclude the individual's ability to successfully and safely complete the study or that may confound study outcomes.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2024-02-02 (Actual); Primary Completion 2024-09-12 (Actual); Study Completion 2024-09-12 (Actual)

PRIMARY OUTCOMES:
To assess the efficacy of the Investigational Product (IP) on Glucose Metabolism as assessed by change in serum fasting glucose levels. | Day 0
  The normal values for normal fasting blood glucose concentration are between 4.11-6.05 mmol/L (74-109 mg/dL).
To assess the efficacy of the Investigational Product (IP) on Glucose Metabolism as assessed by change in serum fasting glucose levels. | Day 90
  The normal values for normal fasting blood glucose concentration are between 4.11-6.05 mmol/L (74-109 mg/dL).

SECONDARY OUTCOMES:
To assess the efficacy of the Investigational Product (IP) on Fat metabolism as assessed by serum lipid profile. | Day 0 and Day 90
  Desirable cholesterol level: < 5.17 mmol/L (< 200 mg/dL); Triglycerides: < 1.70 mmol/L (< 150 mg/dL); HDL Cholesterol - Males: 45 - 65 mg/dL, Females: 35 - 55 mg/dL
To assess the efficacy of the Investigational Product (IP) on future assessment of vitality related biomarkers | Day 0, Day 30 and Day 90
  Blood sample will be collected for post hoc analysis
To assess the efficacy of the Investigational Product (IP) on perceived immune system as assessed by Immune System Questionnaire (ISQ) | Day 0, Day 30, Day 60 and Day 90
  The ISQ has seven questions. The sum score is calculated. Interpretation: 0 = very poor and 10= excellent perceived immune status.
To assess the efficacy of the Investigational Product on Physical energy as assessed by energy VAS | Day 0, Day 14, Day 30, Day 60 and Day 90
  The VAS consists of a 10cm line, with two end points representing 0 ('no energy') and 10 ('most energetic')
To assess the efficacy of the Investigational Product on Fatigue level as assessed by Fatigue Severity Scale (FSS) | Day 0, Day 14, Day 30, Day 60 and Day 90
  The FSS is a self-administered questionnaire with 9 items (questions) investigating the severity of fatigue in different situations during the past week. Grading of each item ranges from 1 to 7, where 1 indicates strong disagreement and 7 indicates strong agreement, and the final score represents the mean value of the 9 items.
To assess the efficacy of the Investigational Product on Sleep as assessed by Pittsburg Sleep Quality Index | Day 0, Day 14, Day 30, Day 60 and Day 90
  In scoring the PSQI, seven component scores are derived, each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality.
To assess the efficacy of the Investigational product on Stress perception as assessed by the Cohen Perceived Stress score | Day 0, Day 14, Day 30, Day 60 and Day 90
  Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress.
  * Scores ranging from 0-13 would be considered low stress.
  * Scores ranging from 14-26 would be considered moderate stress.
  * Scores ranging from 27-40 would be considered high perceived stress.

CONTACTS AND LOCATIONS:
Locations (2):
- India (2):
  - Dr. Khare's Clinic, Mumbai, Maharashtra
  - Dr. Preeti Bawaskar's Clinic, Thane, Maharashtra

IPD SHARING:
Plan to Share IPD: No